CLINICAL TRIAL: NCT03792711
Title: A Controlled, Open-label, Parallel-group, Randomized Study to Evaluate the Effects of Additional Oral Nutritional Supplement With β-hydroxy-β-methylbutyrate on Thigh Muscle Mass in Older People With Pre-frail Status in Taiwan
Brief Title: The Effects of the Oral Nutritional Supplement With β-hydroxy-β-methylbutyrate in Lean Body Mass Among Taiwan Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANTW1701
Record Dates: First submitted 2018-12-11; First posted 2019-01-03 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2019-07

CONDITIONS: Frail Elderly Syndrome; Nutrition Disorders in Old Age; Muscle Loss
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMB group (Experimental): 2 servings (440 mL)/day Ensure® Plus Advance for use as a supplement with or between meals
  Interventions: Dietary Supplement: Ensure® Plus Advance
- Control group (No Intervention): Standard of care includes mainly dietary consultation for healthy aging by dietitians to reach sufficient dietary protein intake.

INTERVENTIONS:
Dietary Supplement: Ensure® Plus Advance — Previous studies suggest that protein supplementation is an effective dietary strategy to decrease frailty by positively influence the weight loss or sarcopenia in elderly.
  Lean body mass includes all body tissue except fat and is well recognized to be associated with an increased risk of morbidity and mortality. Oral nutrition supplements have been shown to increase food intake and body weight, but not lean body mass. In previous studies, β-hydroxy-β-methylbutyrate, which is leucine metabolite, has been shown to enhance protein synthesis and decrease protein degradation leading to increase lean body mass. It showed that β-hydroxy-β-methylbutyrate supplement with exercise increased lean body mass in health elderly population and improved the physical performance in elderly women.
  Arms: HMB group

SUMMARY:
Primary objective:

To evaluate the effects of additional oral nutritional supplement containing β-hydroxy-β-methylbutyrate (HMB) on thigh muscle mass in elderly subjects with pre-frail status

Secondary objectives:

1. To evaluate the effects of additional oral nutritional supplement containing β-hydroxy-β-methylbutyrate on physical performance, nutrition status, and quality of life in elderly subjects with pre-frail status
2. To determine the safety profile of additional oral nutritional supplement containing β-hydroxy-β-methylbutyrate in elderly subjects with pre-frail status

DETAILED DESCRIPTION:
This is a controlled, open-label, parallel-group, randomized, investigator initiated study to evaluate the effectiveness of oral nutritional supplement containing β-hydroxy-β-methylbutyrate (Ensure® Plus Advance) on thigh muscle mass and physical performance in elderly subjects with pre-frail status. The study is planned to enroll a total of 70 elderly subjects with pre-frail status defined by Fried's criteria with modified cutoff values as suggested by Asian Working Group for Sarcopenia (AWGS) for Asian population. The subject to be enrolled will meet the phenotypic definition of pre-frail for one or two of five phenotypic criteria: weakness as measured by grip strength, slow walking speed, low level of physical activity, self-reported exhaustion, and unintentional weight loss.

After obtaining informed consent and the confirmation of eligibility, subjects will be randomized into the HMB or control group in a 1:1 ratio. All enrolled subjects will be under standard care, which is mainly dietary consultation for healthy aging by dietitians to assure sufficient dietary protein intake in all subjects. Subjects assigned to the HMB group will consume 2 bottles of Ensure® Plus Advance per day for 12 weeks additionally, while subjects assigned to the control group will not receive any placebo or active control.

In this study, subjects will be requested for a total of 4 visits at the clinical site, including screening visit, Visit 1 for randomization, Visit 2 at Week 6, and Visit 3 at Week 12 (end of study/EOS). The telephone visit will be scheduled at Week 3 and Week 9 to follow-up with subjects.

Thigh muscle mass of all subjects will be evaluated by MRI. The physical performance of subjects will be determined by short physical performance battery (SPPB) and handgrip strength. The nutrition status of subjects will be measured by MNA® -SF and nutrition biomarkers, including serum albumin, pre-albumin, 25-hydroxy-vitamin D, vitamin B12, and C-reactive protein (CRP). SF-36v2™ Health Survey will be used to evaluate the quality of life of subjects. The safety profile of Ensure® Plus Advance will be determined by monitoring the adverse event (AE/SAE) during the study period. Blood samples of each subject will be collected at Visits 1, 2 and 3 for analysis of nutrition biomarkers. There will be a total of approximately 30 mL of blood to be collected from each subject during the study period.

ELIGIBILITY:
Inclusion Criteria:

Subjects have to meet ALL inclusion criteria to be eligible for participation in the study.

1. Male or female subject with age between 65-80 years old (inclusive)
2. Subject with pre-frail status, which is defined by Fried's criteria
3. Subject who can fully communicate, understand the study, and provide the informed consent

Exclusion Criteria:

Subjects who meet ANY of the following exclusion criteria will be excluded from the study.

1. Subject with BMI > 35 kg/m2
2. Subject with active diseases judged by the investigator as below

   1. Recent stroke (within 6 months prior to screening)
   2. Parkinsonism
   3. Motor neuron disease
   4. Uncontrolled cardiovascular disease
   5. Uncontrolled chronic obstructive pulmonary disease
   6. Chronic kidney disease severe than Stage IIIb
   7. Dementia or other mental illness with cognitive impairment
   8. Uncontrolled depression
   9. Chronic and acute infection
   10. Uncontrolled metabolic diseases including type II diabetes mellitus
   11. Thyroid disease, including hypothyroidism and hyperthyroidism
   12. Uncontrolled gastrointestinal disease (inflammatory bowel disease, Crohn's disease, etc)
3. Subject with a history or evidence of malignancy in the past 5 years (except for non-melanoma skin neoplasia)
4. Subject using any dietary supplementation containing β-hydroxy-β-methylbutyrate within 1 month prior to screening
5. Subject using Ensure® plus Advance within 1 month prior to screening

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
lean body mass | 3 months
  Thigh muscle mass (kg) will be measured by MRI and be further analyzed at Visits 1 and 3 (EOS/ET). The data assessed at Visit 1 will be the baseline. The summary results of thigh muscle mass (kg) at the baseline and subsequent visits, and the change from baseline will be summarized descriptively by groups.
  Changes from baseline within each group will be tested by paired t-test or Wilcoxon signed-rank test with a significance level of 0.05. The change from baseline between groups will be analyzed by two sample t-test or Wilcoxon rank-sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Kung Chen, PhD, Principal Investigator — Institute of Health Policy and Welfare, National Yang-Ming University
Locations (1):
- Taiwan Association of Integrated Care, Taipei, Taiwan